CLINICAL TRIAL: NCT01811407
Title: Impacts of Public Announcements of Goals and Outcomes on Goal Completion
Brief Title: Impacts of Public Announcements of Goals and Outcomes on Goal Completion (Commit to Steps)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Paul J. Resnick, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 9010
Record Dates: First submitted 2013-02-14; First posted 2013-03-14 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Behavior and Behavior Mechanisms
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Private/private (Other): Participants will wear a pedometer for 14-15 weeks and receive a weekly step count target each week. Participants will be required to set a forward-looking commitment each week as to how many days during the following week they will meet their step count target. Commitment and results will be private.
  Interventions: Behavioral: Walking program
- Public/private (Experimental): Participants will wear a pedometer for 14-15 weeks and receive a weekly step count target each week. Commitments are made as in the Private/Private condition. In addition, one Facebook announcement will be posted at the beginning of the week that says how many days the participant thinks they will meet their walking target the following week. An email will also be sent directly to 3 friends the participant chose with the same announcements.
  Interventions: Behavioral: Precommitment announcement; Behavioral: Walking program
- Public/public (Experimental): Participants will wear a pedometer for 14-15 weeks and receive a weekly step count target each week. Commitments will be made as in the Private/Private condition. In addition, one message will be posted to Facebook at the beginning of the week that says how many days the participant thinks they will meet their walking target the following week, and how they did on their previous weekly commitment. An email will also be sent directly to 3 friends the participant chose with the same announcements.
  Interventions: Behavioral: Precommitment announcement; Behavioral: Results announcement; Behavioral: Walking program

INTERVENTIONS:
Behavioral: Precommitment announcement
  Arms: Public/private; Public/public
Behavioral: Results announcement
  Arms: Public/public
Behavioral: Walking program

SUMMARY:
Physical activity is known to help reduce obesity and the problems that accompany it. Walking has many benefits that make it an excellent way for obese people to increase their physical activity. It is hard, however, for people to stick with walking programs. Setting specific and challenging walking targets that are combined with timely feedback about discrepancies between desired and actual performance lead to higher performance. There is conflicting theory and evidence about the effects of publicly announcing those targets on commitment to the targets and on performance.

Our research question is whether public announcements reduce the challenge level of commitments people set, and whether the reputational consequence of public announcements is severe enough to increase performance. The investigators propose a controlled trial that will integrate Facebook with the objective monitoring of walking via the use of pedometers to test the effect of public announcements on commitments and step counts.

All participants will wear a pedometer and upload via the internet for 14 to 15 weeks, depending on their date of randomization. The first 2 to 3 weeks the investigators will determine the participant's baseline step counts. The following 12 weeks, the investigators will recommend a daily step count target based on the median number of steps the participants walked the previous week. Each week, participants will set a commitment by stating the number of days in the following week that he/she will meet the computer-set step count target.

Commitments will be entered into an interface that will link with Facebook. Participants will select who of their Facebook friends will receive their commitments and/or results via Facebook posts. The interface will distribute those posts in a way that fits in with existing online social practices.

There will be 3 experimental conditions. 1.) No public announcements 2.) Public announcement of commitment and 3.) Public announcement of commitment and results. In addition, groups 2 and 3 will provide us with emails of 3 friends or family members who will act as the participant's support team. The investigators will send announcements directly to support team members.

The investigators plan to recruit 165 participants primarily by obtaining lists of potentially eligible University of Michigan Health System patients from the clinical data repository, and sending targeted letters to these patients. Because this research - and the physical activity programs it will inform - aims to reach a large number of people efficiently, enrollment will take place online with a click-through consent document. The investigators have extensive experience with delivering online walking programs in similar populations.

The investigators hope to learn best practices for using public announcements and online social networks to encourage people to exercise more or to otherwise promote wellness.

ELIGIBILITY:
Inclusion Criteria

* Has received treatment from a UMHS provider within the previous 6 months.
* BMI ≥ 30
* Age ≥ 18
* Must be sedentary, defined by less than 150 minutes of self-reported activity per week.
* Must have access to a computer with an Internet connection that can accept USB uploads.
* Must have a Facebook account and have at least 50 friends on it.
* Must be able to communicate in English.

Exclusion Criteria

* Currently pregnant
* Unable to comfortably walk at least a block without the assistance of a cane or walker.
* Not competent to sign a consent form.
* Absolute or relative contraindications to walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The number of days the participant met the weekly step count target. | Participants will be followed for 14 to 15 weeks, depending on the date of randomization.

SECONDARY OUTCOMES:
The number of days the participants committed to walking. | Participants will be followed for 14 to 15 weeks, depending on the date of randomization.
The change in step counts from baseline. | Participants will be followed for 14 to 15 weeks, depending on the date of randomization.
The number of days the participants wore the pedometer. | Participants will be followed for 14 to 15 weeks, depending on the date of randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Resnick, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States